CLINICAL TRIAL: NCT07176403
Title: Effect of Intradialytic Exercise Program on Sleep Quality, Depression and Anxiety in Hemodialysis Patients
Brief Title: Effect of Intradialytic Exercise on Sleep, Depression and Anxiety in HD Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Mohamed Mamdouh Mahmoud Mohamed Elsayed , MD, Associate professor, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: exercise effect on HD patients
Record Dates: First submitted 2025-09-09; First posted 2025-09-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Intradialytic Exercise
Keywords: Intradialytic exercise; sleep; depression; anxiety; hemodialysis
MeSH Terms: conditions — Depression; Anxiety Disorders | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: The study will include seventy patients maintained on regular hemodialysis in Alexandria University Hospitals.
  Patients will be divided into two groups:
  Group (A): 50 patients will perform exercise during hemodialysis session. Group (B): 50 patients will not be assigned to any exercise program (as a control group).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise group (Experimental): 50 patients will undergo Exercise training program for twelve weeks during hemodialysis session.
  1. Type of exercise: aerobic exercise training sessions using a lower limb ergometer.
  2. Frequency: three times per week.
  3. Duration: thirty minutes per session.
  Interventions: Other: intradialytic exercise
- control group (Placebo Comparator): 50 patients will not perform exercise during hemodialysis session
  Interventions: Other: control group

INTERVENTIONS:
Other: intradialytic exercise — 50 patients will undergo Exercise training program for twelve weeks during hemodialysis session.
  1. Type of exercise: aerobic exercise training sessions using a lower limb ergometer.
  2. Frequency: three times per week.
  3. Duration: thirty minutes per session.
  Arms: Exercise group
Other: control group — 50 patients will not perform exercise during hemodialysis session
  Arms: control group

SUMMARY:
this study aims To assess the effect of intradialytic exercise program on sleep quality, depression and anxiety in HD Patients.

DETAILED DESCRIPTION:
Intradialytic exercise is a common recommendation given to encourage patients to be physically active. Previous studies have suggested that intradialytic exercise is effective in reducing fatigue severity, improving sleep quality, enhancing exercise tolerance, improving quality of life and even psychological status. Research also revealed that intradialytic exercise can increase the efficacy of dialysis, subsequently alleviating inflammation, improving nutrition and bone mineral density. Patients typically undergo two or three hemodialysis sessions a week, with each session lasting for approximately 4 hours. Since many patients maintain bed rest during HD sessions, intradialytic exercise can be a potentially useful approach to improve their health without consuming extra time during the interdialytic period.

ELIGIBILITY:
Inclusion Criteria:

1. ESKD patients on maintenance hemodialysis for more than three months.
2. Age more than 18 years.

Exclusion Criteria:

1. Mentally or physically unfit patients or with severe psychiatric illness.
2. Patients who receive any psychotropic medications.
3. Patients with overt ischemic heart disease or cardiac decompensation.
4. Anemic patients (Hb ≤ 8 mg/dl).
5. Patients presented with severe bone pains or muscle weakness secondary to chronic kidney disease-mineral and bone disorder (CKD-MBD).
6. Patients with advanced lower limbs joints disease.
7. Lower limb amputation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-07-15 (Actual); Primary Completion 2025-10-15 (Estimated); Study Completion 2025-11-15 (Estimated)

PRIMARY OUTCOMES:
change in sleep quality | 12 weeks
  by using The Pittsburgh sleep Quality Index (PSQI).
change in depression scale | 12 weeks
  by using Beck Depression inventory (BDI)
change in anxiety level | 12 weeks
  by using The Beck Anxiety Inventory (BAI) scoring

SECONDARY OUTCOMES:
effect on dialysis adequacy | 12 weeks
  by assessing urea reduction ratio (URR)
effect on lipid profile | 12 weeks
  by assessing triglycerides and cholesterol

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed mamdouh Elsayed, MD, Principal Investigator — Associate professor; Iman Ezzat Elgohary, MD, Principal Investigator — professor; Marwa Mohamed Hassan, MD, Study Chair — professor; Heba Essam Abou EL wafa, MD, Study Chair — professor; Raghda Ashraf AboTawila, MBBCh, Study Chair — resident
Locations (1):
- Faculty of Medicine, Aexandria University, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Jung TD, Park SH. Intradialytic exercise programs for hemodialysis patients. Chonnam Med J. 2011 Aug;47(2):61-5. doi: 10.4068/cmj.2011.47.2.61. Epub 2011 Aug 31. PMID 22111062
- [Background] Rajan EJ, Subramanian S. The effect of depression and anxiety on the performance status of end-stage renal disease patients undergoing hemodialysis. Saudi J Kidney Dis Transpl. 2016 Mar;27(2):331-4. doi: 10.4103/1319-2442.178555. PMID 26997387
- [Background] Mollayeva T, Thurairajah P, Burton K, Mollayeva S, Shapiro CM, Colantonio A. The Pittsburgh sleep quality index as a screening tool for sleep dysfunction in clinical and non-clinical samples: A systematic review and meta-analysis. Sleep Med Rev. 2016 Feb;25:52-73. doi: 10.1016/j.smrv.2015.01.009. Epub 2015 Feb 17. PMID 26163057
- [Background] Gordon L, McGrowder DA, Pena YT, Cabrera E, Lawrence-Wright M. Effect of exercise therapy on lipid parameters in patients with end-stage renal disease on hemodialysis. J Lab Physicians. 2012 Jan;4(1):17-23. doi: 10.4103/0974-2727.98665. PMID 22923917